CLINICAL TRIAL: NCT00541931
Title: Pilot Investigation of a Multinutrient Supplement on Skin Aging and Aging Metabolites in Healthy Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Nu Skin Enterprises (Industry)
Responsible Party: Principal Investigator, Anne Chang, Professor, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10622
Record Dates: First submitted 2007-10-05; First posted 2007-10-10 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Skin Diseases
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nonsmoker (Other): Nonsmokers Intervention: Dietary Supplement: LifePak Nano
  Interventions: Drug: Dietary Supplement: LifePak Nano
- Smoker (Other): Smoker arm Intervention: Dietary Supplement: LifePak Nano
  Interventions: Drug: Dietary Supplement: LifePak Nano

INTERVENTIONS:
Drug: Dietary Supplement: LifePak Nano — Daily use
  Other Names: Life Pak Nano

SUMMARY:
We are seeking healthy female volunteers to determine if multinutrient supplementation affects visible signs of skin aging as well as blood measurements of aging. We are seeking smokers and non-smokers.

DETAILED DESCRIPTION:
Skin antioxidant levels as well as blood metabolites may change as the human body ages1,2. Although the chronological aging process is unstoppable, the physical signs of aging, particularly characteristics of the skin, may be delayed through a variety of medical interventions such as topical medications or resurfacing lasers. It is not currently known whether skin carotenoid antioxidant levels correlate with skin aging characteristics, although studies with other antioxidants suggest this may be true 3. In addition, while selected blood metabolites correlate with changes in age2, we do not know if this correlates with skin changes. Our current study focuses on whether differences in skin carotenoid levels and blood metabolite levels correlate with skin aging characteristics in age-matched subjects. Furthermore, we will explore whether three months consumption with a commercial multi-nutrient formulation (LifePak Nano) affects metabolic markers of aging, skin aging characteristics including skin elasticity and transepidermal water loss. We will also examine whether smokers respond differently from nonsmokers in the above parameters after supplementation.

ELIGIBILITY:
Inclusion Criteria:- Fitzpatrick Skin type I or II

* Nonpregnant Females, age 18-30 or 50-70
* Body Mass Index Normal or Overweight
* If age 18-30, must be non-smoker
* Willing to fast for 8 hours prior to a blood draw; Exclusion Criteria:- History of cosmetic surgery
* Use of anti-aging medications within 3 months of enrollment
* Use of over-the-counter anti-aging creams (not sunscreens) more than once per week within one month of enrollment
* Use of dietary supplements including vitamins within one month of enrollment
* Use of tanning beds or excessive UV exposure (greater than 2 hours per day) within one month of enrollment
* Use of sunless tanners within one month of enrollment
* Uncontrolled or ongoing serious medical condition
* Participation in another clinical study involving use of an investigational drug or product
* Medical condition which, at the discretion of the investigator, will have a significant impact on ability to judge participant's skin characteristics, including age.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-10; Primary Completion 2008-03 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Anne Lynn S. Chang, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Spitale RC, Cheng MY, Chun KA, Gorell ES, Munoz CA, Kern DG, Wood SM, Knaggs HE, Wulff J, Beebe KD, Chang AL. Differential effects of dietary supplements on metabolomic profile of smokers versus non-smokers. Genome Med. 2012 Feb 23;4(2):14. doi: 10.1186/gm313. PMID 22360970

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy female volunteers in the community aged >50 years
Groups:
- Nonsmoker: Nonsmokers Intervention: Dietary Supplement: LifePak Nano
  Dietary Supplement: LifePak Nano : Daily use
- Smoker: Smoker arm Intervention: Dietary Supplement: LifePak Nano
  Dietary Supplement: LifePak Nano : Daily use
Period: Overall Study
Arm/Group | Nonsmoker | Smoker
Started | 22 | 15
Completed | 17 | 11
Not Completed | 5 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Transportation Issue | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants completing the protocol were included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nonsmoker | Smoker | Total
Number analyzed (Participants) | 17 | 11 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 11 | 28
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (6.3) | 56.3 (5.0) | 56.0 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 28
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 11 | 28
Fine wrinkling as assessed by clinician [Mean (Standard Deviation); unit: units on a scale] — Population: Assessed by 4 dermatologists blinded to chronological age and smoking status, on a 10-point Likert scale (min 1/max 10); lower scores indicate less wrinkling and higher scores indicate more wrinkling. Values are the average of scores given by the four raters.
  units on a scale | 8.35 (1.80) | 8.70 (1.70) | 8.37 (1.75)

OUTCOME MEASURES:

1. Primary Outcome: Fold Change in Long Chain Fatty Acids
Description: Peripheral blood long chain fatty acids were measured. Fold change of 1 = no difference; if metabolites decrease at week 12 from baseline, the fold change will be <1.
Time Frame: Baseline; Week 12
Population: Participants completing the protocol were included in the analysis.
Measure: Mean (Full Range); unit: Fold Change in long chain fatty acids
Arm/Group | Nonsmoker | Smoker
Number analyzed (Participants) | 17 | 11
Fold Change in long chain fatty acids | 1 [0 to 1] | 0.76 [0 to 1]

2. Primary Outcome: Change in Fine Wrinkling
Description: Assessed by 4 dermatologists blinded to chronological age and smoking status, on a 10-point Likert scale (min 1/max 10); lower scores indicate less wrinkling and higher scores indicate more wrinkling. Values are the average of scores given by the four raters. Change was calculated as the baseline value minus the week 12 value.
Time Frame: Baseline; week 12
Population: Participants completing the protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nonsmoker | Smoker
Number analyzed (Participants) | 17 | 11
units on a scale | 0.24 (1.82) | -1.77 (2.74)

ADVERSE EVENTS:
Time Frame: Duration of enrollee participation (12 weeks)
Description: All study participants were asked about adverse events at every study visit with results graded and recorded
Arm/Group | Nonsmoker | Smoker
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/15
Other Adverse Events (participants affected / at risk) | 14/22 | 6/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nonsmoker (N=22) | Smoker (N=15)
Body Aches (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Headaches (Nervous system disorders) | 11 (11) | 3 (3)

LIMITATIONS AND CAVEATS:
Sample size limitation, short term nature of study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No